CLINICAL TRIAL: NCT01491243
Title: Neutrophil gElatinase-associated Lipocalin alloWs Intensive treatMent Of cOntrast Induced Nephropathy in Patients With Urgent/Emergency Percutaneous Coronary Intervention
Brief Title: N-GAL Allows Intensive Treatment of Contrast Induced Nephropathy
Acronym: NEW-MOON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 652/2011/D
Record Dates: First submitted 2011-12-11; First posted 2011-12-13 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: contrast-induced nephropathy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive treatment group (Active Comparator): Patients will receive high concentration sodium bicarbonate (3 ml/kg/h for 1 hour, then 1 ml/kg/h for 7 h) followed by i.v. saline for 48 h after PCI in case of abnormal NGAL findings
  Interventions: Drug: Intensive treatment with sodium bicarbonate
- Standard treament group (Active Comparator): Patients will receive i.v. 1 ml/kg/h saline infusion for 48 h after PCI in case of abnormal NGAL findings
  Interventions: Drug: Standard treatment with saline infusion

INTERVENTIONS:
Drug: Intensive treatment with sodium bicarbonate — i.v., sodium bicarbonate (3 ml/kg/h for 1 hour, then 1 ml/kg/h for 7 h) followed by i.v. saline for 48 h in case of abnormal NGAL findings
  Arms: Intensive treatment group
Drug: Standard treatment with saline infusion — i.v. 1 ml/kg/h saline infusion for 48 h in case of abnormal NGAL findings
  Arms: Standard treament group

SUMMARY:
Patients who undergo urgent/emergency coronary angiography can not receive any preventive treatment of contrast induced nephropathy. We tested the hypothesis that Neutrophil gelatinase-associated lipocalin (NGAL), a new biomarker predictive for AKI, allows early and effective treatment of contrast induced nephropathy in patients with urgent/emergency coronary angiography

DETAILED DESCRIPTION:
Background Patients who undergo urgent/emergency coronary angiography can not receive any preventive treatment of contrast induced nephropathy.

An acute kidney injury is generally detected too late to allow effective intervention in patients who undergo urgent/emergency coronary angiography.

Neutrophil gelatinase-associated lipocalin (NGAL) is a new biomarker predictive for AKI already shown to be useful for earlier diagnosis of contrast induced nephropathy.

Purpose The primary objective of this study is to to test the hypothesis that a NGAL-driven early intensive strategy can reduce the occurrence of contrast induced nephropathy in patients with urgent/emergency coronary angiography

ELIGIBILITY:
Inclusion Criteria:

* Indication to urgent/emergency coronary angiography
* Normal renal function (eGFR> 60 ml/min/1.73 m2)
* Moderate or high Mehran's risk score for CIN (>11).
* Able to understand and willing to sign the informed consent form

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of contrast induced nephropathy | Baseline and 48 hours after angiography
  Absolute increase in serum creatinine equal to or greater than 0.5 mg/dL detected 48 hours after angiography as compared with baseline value

SECONDARY OUTCOMES:
Post-angiographic changes in renal function parameters | Baseline and 48 hours after angiography
  Changes in creatinine levels and estimated glomerular filtration rate at 48-hour evaluation after angiography as compared with baseline values

CONTACTS AND LOCATIONS:
Locations (1):
- University La Sapienza, Rome, Italy